CLINICAL TRIAL: NCT00192127
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety of a Bivalent Vaccine of New 6:2 Influenza Virus Reassortants in Healthy Adults
Brief Title: Study to Evaluate the Safety of a Bivalent Vaccine of New 6:2 Influenza Virus Reassortants in Healthy Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Robert Walker, M.D., MedImmune Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MI-CP113
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-12-18 (Estimated); Status verified 2007-12

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — FluMist

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator): FluMist
  Interventions: Biological: FluMist
- 2 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: FluMist — A single dose of either bivalent vaccine or placebo mist by intranasal spray on Study Day 0.
  Arms: 1
Other: Placebo — A single dose of either bivalent vaccine or placebo mist by intranasal spray on Study Day 0
  Arms: 2

SUMMARY:
This study is to assess the safety of a bivalent vaccine of two new 6:2 influenza virus reassortants in healthy adults prior to the release of the trivalent vaccine (FluMist) containing them.

DETAILED DESCRIPTION:
The primary study objective is to assess the safety of a bivalent vaccine of two new 6:2 influenza virus reassortants in healthy adults prior to the release of the trivalent vaccine (FluMist) containing them. Safety will be demonstrated by similar fever rates (oral temperature ≥101°F Days 0-7) in vaccine and placebo recipients.

ELIGIBILITY:
Inclusion Criteria:

* 18-49 years of age (not yet reached their 50th birthday);
* In good health;
* Available by telephone;
* Ability to understand and comply with the requirements of the protocol; and
* Signed informed consent and HIPAA authorization.

Exclusion Criteria:

* Any condition for which the inactivated influenza vaccine is indicated, including: chronic disorders of the pulmonary or cardiovascular systems, including asthma; chronic metabolic diseases (including diabetes mellitus) renal dysfunction, or hemoglobinopathies which required regular medical follow-up or hospitalization during the preceding year;
* Acute febrile (>100.0°F oral) and/or respiratory illness, including cough or sore throat, within the 14 days prior to enrollment;
* Hypersensitivity to egg or egg protein;
* Hypersensitivity to gentamicin;
* Any known immunosuppressive condition or immune deficiency disease, including HIV infection, or ongoing immunosuppressive therapy;
* History of Guillan-Barré Syndrome;
* Household contact who is immunocompromised (participant should also avoid close contact with immunocompromised individuals for at least 21 days);
* Participation in another investigational trial within 30 days prior to enrollment or expected enrollment in another investigational trial during this study;
* Chronic or regular use of antipyretic or analgesic medication on a daily or every other day basis; Notes: A daily dose of 81 mg of aspirin is not considered a contraindication to enrollment. Discontinuation of prophylactic use of antipyretic or analgesic medications at the time of enrollment and for fourteen days following vaccination is not considered a contraindication to enrollment.
* Pregnancy or, in biologically capable women (e.g., menses within the last year) participant does not agree to use acceptable birth control measures as determined by the investigator continuously for three months after enrolling into the study (for those biologically capable, a urine pregnancy test must be performed on the day of vaccination with a negative result);
* Breastfeeding or lactating women;
* Administration of intranasal medications within two weeks prior to enrollment or expected receipt during this study;
* Employees of the investigational site or their family member or any individuals involved with the conduct of the study; and
* Any condition that in the opinion of the investigator, might interfere with the vaccine evaluation.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300
Dates: Start 2004-08; Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study is fever (Day 0-7) defined as oral temperature ³101°F. | Day 0-7

SECONDARY OUTCOMES:
Secondary endpoints of the study include other reported reactogenicity events and other adverse events that occur within seven days (Day 0-7) and fourteen days (Day 0-14) following vaccination | Days 0-7; 0-14

CONTACTS AND LOCATIONS:
Overall Officials: Robert Walker, MD, Study Director — Sponsor GmbH
Locations (1):
- SFBC International, Inc, Miami, Florida, United States